CLINICAL TRIAL: NCT01589367
Title: Phase II Randomized Study of Neoadjuvant Metformin Plus Letrozole vs Placebo Plus Letrozole for ER-positive Postmenopausal Breast Cancer
Brief Title: Neoadjuvant Letrozole Plus Metformin vs Letrozole Plus Placebo for ER-positive Postmenopausal Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KBCSG 013
Record Dates: First submitted 2012-04-17; First posted 2012-05-01 (Estimated); Last update posted 2018-09-10 (Actual); Status verified 2017-06

CONDITIONS: Hormone Receptor Positive Malignant Neoplasm of Breast
Keywords: neoadjuvant endocrine therapy; metformin; postmenopausal breast cancer
MeSH Terms: interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm1_ Metformin (Experimental): Letrozole with concurrent metformin
  Interventions: Drug: Metformin
- Arm 2_ Letrole alone (Placebo Comparator): Letrozole with placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Metformin — Metformin HCl 500mg(morning/evening) PO daily x 1week Metformin HCl 1000mg(morning)and 500mg(evening)PO daily x 1week Metformin HCl 1000mg(morning/evening) PO daily x 22weeks
  Other Names: Arm1_Metformin_experimental
  Arms: Arm1_ Metformin
Drug: Placebo — Letrozole 2.5mg PO daily + Placebo 1 tablet PO 2/day x 1week Letrozole 2.5mg PO daily + Placebo 2 tablet+ 1 tablet PO x 1 week Letrozole 2.5mg PO daily + Placebo 2 tablet PO 2/day x 22 weeks
  Other Names: Arm2_Letrozole alone_Placebo
  Arms: Arm 2_ Letrole alone

SUMMARY:
Preoperative letrozole versus letrozole with metformin in postmenopausal Estrogen receptor positive breast cancer patients

Phase II multicenter 1:1 randomized clinical trial Total 208 patients

Primary endpoint Clinical response rate

Secondary endpoint Pathologic complete response rate Breast conserving surgery rate Percent mammographic density change Ki67(%) change after 4week medication of 2nd core needle biopsy Toxicity profile of neoadjuvant letrozole, metformin

DETAILED DESCRIPTION:
To identify the anti-tumor effect of metformin with preoperatively given letrozole in postmenopausal estrogen receptor positive breast cancer patients

ELIGIBILITY:
Inclusion Criteria:

* Estrogen receptor positive breast cancer
* Clinically measurable tumor size(stage II/III)
* No evidence of distant metastasis
* Postmenopause women 'Age≥60yr' OR 'previous bilateral oophorectomy' OR 'FSH>30 with no bleeding history within 1yr'
* ECOG 0-2
* Adequate hepatorenal, bone marrow function 'serum Cr<1.4mg/dL' AND 'Bilirubin< upper limit of normal x 1.5 AND 'AST/ALT < upper limit of normal x 1.8 AND 'ALP < upper limit of normal x 1.8 AND 'Hemoglobin >10 g/dL' AND 'ANC >1,500/mm3' AND 'Platelet >100,000/mm3'
* Spontaneous signed into the written informed consent

Exclusion Criteria:

* Who does not meet the above inclusion criteria
* History of other carcinoma
* Uncontrolled infection
* History of psychiatric, epileptic disease
* Male breast cancer
* Diabetes 'HbA1c≥6.5' OR 'FBS≥126mg/dL'
* Hypersensitivity or intolerance to metformin
* Risk of metformin associated lactic acidosis 'Congestive heart disease of NYHA Class llll/IV' OR 'History of other acidosis' OR 'Alcohol intake more than either 3 bottles beer OR 1 bottle Soju'
* During medication of metformin, sulfonylureas, thiazolidinediones, insulin
* Diffuse microcalcification in mammogram
* Multiple OR bilateral OR inflammatory breast cancer
* Chemotherapy or endocrine therapy within 2yr due to history of breast cancer

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2012-05; Primary Completion 2018-04 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Clinical response rate | 24week(after completing medication, preoperatively)
  Comparing with RECIST 1.1 From baseline to 24week(after completing medication, preoperatively)

SECONDARY OUTCOMES:
Pathologic complete response rate | Postoperation(within 26weeks after starting medication)
  In case that under postoperative biopsy, residual breast cancer cell is not present in primary lesion and lymph node.
Changes of Ki67(%) | Baseline-4week(second core needle biopsy)
  IHC is performed for formalin-fixed paraffin embedded tissue at the central laboratory. Ki67 is recorded as % and percentage reduction of baseline and Ki67 expressed cell on day28 are compared.
Breast conservation rate | Baseline-postoperation(within 26weeks after starting medication)
  Before pre-operative anti hormone therapy, the patients are classified into following three types
  1. Candidate for BCS
  2. Marginal for breast conservation surgery
  3. Candidate for mastectomy only
  4. Inoperable by standard mastectomy Classification of each type shall be determined by each researcher of each institution subjectively. For future separate objective analysis, central institution will collect image file of mammography of each patient.
  Type of operation being actually performed in each type is compared. (BCS vs mastectomy)
Breast density change | Baseline-24week(after completing medication, preoperatively)
  Percent mammographic density (%) of cranial-caudal view of opposite breast is measured/compared based on continued variable by using validated computer-assisted thresholding program called Cumulus software (University Toronto, Toronto, Ontario, Canada).
Toxicity profile of letrozole and metformin | throughout the study
  based on NCI-CTCAE version 4.0

CONTACTS AND LOCATIONS:
Overall Officials: Wonshik Han, MD PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Fisher B, Bryant J, Wolmark N, Mamounas E, Brown A, Fisher ER, Wickerham DL, Begovic M, DeCillis A, Robidoux A, Margolese RG, Cruz AB Jr, Hoehn JL, Lees AW, Dimitrov NV, Bear HD. Effect of preoperative chemotherapy on the outcome of women with operable breast cancer. J Clin Oncol. 1998 Aug;16(8):2672-85. doi: 10.1200/JCO.1998.16.8.2672. PMID 9704717
- [Background] Wolmark N, Wang J, Mamounas E, Bryant J, Fisher B. Preoperative chemotherapy in patients with operable breast cancer: nine-year results from National Surgical Adjuvant Breast and Bowel Project B-18. J Natl Cancer Inst Monogr. 2001;(30):96-102. doi: 10.1093/oxfordjournals.jncimonographs.a003469. PMID 11773300
- [Background] van der Hage JA, van de Velde CJ, Julien JP, Tubiana-Hulin M, Vandervelden C, Duchateau L. Preoperative chemotherapy in primary operable breast cancer: results from the European Organization for Research and Treatment of Cancer trial 10902. J Clin Oncol. 2001 Nov 15;19(22):4224-37. doi: 10.1200/JCO.2001.19.22.4224. PMID 11709566
- [Background] Toi M, Nakamura S, Kuroi K, Iwata H, Ohno S, Masuda N, Kusama M, Yamazaki K, Hisamatsu K, Sato Y, Kashiwaba M, Kaise H, Kurosumi M, Tsuda H, Akiyama F, Ohashi Y, Takatsuka Y; Japan Breast Cancer Research Group (JBCRG). Phase II study of preoperative sequential FEC and docetaxel predicts of pathological response and disease free survival. Breast Cancer Res Treat. 2008 Aug;110(3):531-9. doi: 10.1007/s10549-007-9744-z. Epub 2007 Sep 19. PMID 17879158
- [Background] Guarneri V, Broglio K, Kau SW, Cristofanilli M, Buzdar AU, Valero V, Buchholz T, Meric F, Middleton L, Hortobagyi GN, Gonzalez-Angulo AM. Prognostic value of pathologic complete response after primary chemotherapy in relation to hormone receptor status and other factors. J Clin Oncol. 2006 Mar 1;24(7):1037-44. doi: 10.1200/JCO.2005.02.6914. PMID 16505422
- [Background] Aapro M, Monfardini S, Jirillo A, Basso U. Management of primary and advanced breast cancer in older unfit patients (medical treatment). Cancer Treat Rev. 2009 Oct;35(6):503-8. doi: 10.1016/j.ctrv.2009.04.002. Epub 2009 Sep 16. PMID 19762156
- [Background] Eiermann W, Paepke S, Appfelstaedt J, Llombart-Cussac A, Eremin J, Vinholes J, Mauriac L, Ellis M, Lassus M, Chaudri-Ross HA, Dugan M, Borgs M; Letrozole Neo-Adjuvant Breast Cancer Study Group. Preoperative treatment of postmenopausal breast cancer patients with letrozole: A randomized double-blind multicenter study. Ann Oncol. 2001 Nov;12(11):1527-32. doi: 10.1023/a:1013128213451. PMID 11822750
- [Background] Mlineritsch B, Tausch C, Singer C, Luschin-Ebengreuth G, Jakesz R, Ploner F, Stierer M, Melbinger E, Menzel C, Urbania A, Fridrik M, Steger G, Wohlmuth P, Gnant M, Greil R; Austrian Breast, Colorectal Cancer Study Group (ABCSG). Exemestane as primary systemic treatment for hormone receptor positive post-menopausal breast cancer patients: a phase II trial of the Austrian Breast and Colorectal Cancer Study Group (ABCSG-17). Breast Cancer Res Treat. 2008 Nov;112(1):203-13. doi: 10.1007/s10549-007-9843-x. Epub 2007 Dec 22. PMID 18158620
- [Background] Semiglazov VF, Semiglazov VV, Dashyan GA, Ziltsova EK, Ivanov VG, Bozhok AA, Melnikova OA, Paltuev RM, Kletzel A, Berstein LM. Phase 2 randomized trial of primary endocrine therapy versus chemotherapy in postmenopausal patients with estrogen receptor-positive breast cancer. Cancer. 2007 Jul 15;110(2):244-54. doi: 10.1002/cncr.22789. PMID 17538978
- [Background] Ben Sahra I, Laurent K, Loubat A, Giorgetti-Peraldi S, Colosetti P, Auberger P, Tanti JF, Le Marchand-Brustel Y, Bost F. The antidiabetic drug metformin exerts an antitumoral effect in vitro and in vivo through a decrease of cyclin D1 level. Oncogene. 2008 Jun 5;27(25):3576-86. doi: 10.1038/sj.onc.1211024. Epub 2008 Jan 21. PMID 18212742
- [Background] Bowker SL, Majumdar SR, Veugelers P, Johnson JA. Increased cancer-related mortality for patients with type 2 diabetes who use sulfonylureas or insulin: Response to Farooki and Schneider. Diabetes Care. 2006 Aug;29(8):1990-1. doi: 10.2337/dc06-0997. No abstract available. PMID 16873829
- [Background] Evans JM, Donnelly LA, Emslie-Smith AM, Alessi DR, Morris AD. Metformin and reduced risk of cancer in diabetic patients. BMJ. 2005 Jun 4;330(7503):1304-5. doi: 10.1136/bmj.38415.708634.F7. Epub 2005 Apr 22. No abstract available. PMID 15849206
- [Background] Guppy A, Jamal-Hanjani M, Pickering L. Anticancer effects of metformin and its potential use as a therapeutic agent for breast cancer. Future Oncol. 2011 Jun;7(6):727-36. doi: 10.2217/fon.11.49. PMID 21675836
- [Background] Garcia A, Tisman G. Metformin, B(12), and enhanced breast cancer response to chemotherapy. J Clin Oncol. 2010 Jan 10;28(2):e19; author reply e20. doi: 10.1200/JCO.2009.25.7857. Epub 2009 Nov 30. No abstract available. PMID 19949002
- [Background] Jiralerspong S, Palla SL, Giordano SH, Meric-Bernstam F, Liedtke C, Barnett CM, Hsu L, Hung MC, Hortobagyi GN, Gonzalez-Angulo AM. Metformin and pathologic complete responses to neoadjuvant chemotherapy in diabetic patients with breast cancer. J Clin Oncol. 2009 Jul 10;27(20):3297-302. doi: 10.1200/JCO.2009.19.6410. Epub 2009 Jun 1. PMID 19487376
- [Background] Martin-Castillo B, Dorca J, Vazquez-Martin A, Oliveras-Ferraros C, Lopez-Bonet E, Garcia M, Del Barco S, Menendez JA. Incorporating the antidiabetic drug metformin in HER2-positive breast cancer treated with neo-adjuvant chemotherapy and trastuzumab: an ongoing clinical-translational research experience at the Catalan Institute of Oncology. Ann Oncol. 2010 Jan;21(1):187-9. doi: 10.1093/annonc/mdp494. Epub 2009 Nov 2. No abstract available. PMID 19884247
- [Background] Baselga J, Semiglazov V, van Dam P, Manikhas A, Bellet M, Mayordomo J, Campone M, Kubista E, Greil R, Bianchi G, Steinseifer J, Molloy B, Tokaji E, Gardner H, Phillips P, Stumm M, Lane HA, Dixon JM, Jonat W, Rugo HS. Phase II randomized study of neoadjuvant everolimus plus letrozole compared with placebo plus letrozole in patients with estrogen receptor-positive breast cancer. J Clin Oncol. 2009 Jun 1;27(16):2630-7. doi: 10.1200/JCO.2008.18.8391. Epub 2009 Apr 20. PMID 19380449
- [Background] Hadad S, Iwamoto T, Jordan L, Purdie C, Bray S, Baker L, Jellema G, Deharo S, Hardie DG, Pusztai L, Moulder-Thompson S, Dewar JA, Thompson AM. Evidence for biological effects of metformin in operable breast cancer: a pre-operative, window-of-opportunity, randomized trial. Breast Cancer Res Treat. 2011 Aug;128(3):783-94. doi: 10.1007/s10549-011-1612-1. Epub 2011 Jun 8. PMID 21655990
- [Background] Brown KA, Hunger NI, Docanto M, Simpson ER. Metformin inhibits aromatase expression in human breast adipose stromal cells via stimulation of AMP-activated protein kinase. Breast Cancer Res Treat. 2010 Sep;123(2):591-6. doi: 10.1007/s10549-010-0834-y. Epub 2010 Mar 19. PMID 20300828
- [Background] Takemura Y, Osuga Y, Yoshino O, Hasegawa A, Hirata T, Hirota Y, Nose E, Morimoto C, Harada M, Koga K, Tajima T, Yano T, Taketani Y. Metformin suppresses interleukin (IL)-1beta-induced IL-8 production, aromatase activation, and proliferation of endometriotic stromal cells. J Clin Endocrinol Metab. 2007 Aug;92(8):3213-8. doi: 10.1210/jc.2006-2486. Epub 2007 May 15. PMID 17504902
- [Background] Abu Hashim H, Shokeir T, Badawy A. RETRACTED: Letrozole versus combined metformin and clomiphene citrate for ovulation induction in clomiphene-resistant women with polycystic ovary syndrome: a randomized controlled trial. Fertil Steril. 2010 Sep;94(4):1405-1409. doi: 10.1016/j.fertnstert.2009.07.985. Epub 2009 Sep 3. PMID 19732888
- [Background] Goodwin PJ, Pritchard KI, Ennis M, Clemons M, Graham M, Fantus IG. Insulin-lowering effects of metformin in women with early breast cancer. Clin Breast Cancer. 2008 Dec;8(6):501-5. doi: 10.3816/CBC.2008.n.060. PMID 19073504
- [Background] Goldenberg N, Glueck CJ, Loftspring M, Sherman A, Wang P. Metformin-diet benefits in women with polycystic ovary syndrome in the bottom and top quintiles for insulin resistance. Metabolism. 2005 Jan;54(1):113-21. doi: 10.1016/j.metabol.2004.08.007. PMID 15562389
- [Background] Romualdi D, Costantini B, Selvaggi L, Giuliani M, Cristello F, Macri F, Bompiani A, Lanzone A, Guido M. Metformin improves endothelial function in normoinsulinemic PCOS patients: a new prospective. Hum Reprod. 2008 Sep;23(9):2127-33. doi: 10.1093/humrep/den230. Epub 2008 Jun 20. PMID 18567896
- [Background] Baillargeon JP, Jakubowicz DJ, Iuorno MJ, Jakubowicz S, Nestler JE. Effects of metformin and rosiglitazone, alone and in combination, in nonobese women with polycystic ovary syndrome and normal indices of insulin sensitivity. Fertil Steril. 2004 Oct;82(4):893-902. doi: 10.1016/j.fertnstert.2004.02.127. PMID 15482765
- [Background] Ou HY, Cheng JT, Yu EH, Wu TJ. Metformin increases insulin sensitivity and plasma beta-endorphin in human subjects. Horm Metab Res. 2006 Feb;38(2):106-11. doi: 10.1055/s-2006-925128. PMID 16523411
- [Background] Tankova T, Dakovska L, Kirilov G, Koev D. Metformin in the treatment of obesity in subjects with normal glucose tolerance. Rom J Intern Med. 2003;41(3):269-75. PMID 15526510
- [Background] Anisimov VN, Berstein LM, Egormin PA, Piskunova TS, Popovich IG, Zabezhinski MA, Kovalenko IG, Poroshina TE, Semenchenko AV, Provinciali M, Re F, Franceschi C. Effect of metformin on life span and on the development of spontaneous mammary tumors in HER-2/neu transgenic mice. Exp Gerontol. 2005 Aug-Sep;40(8-9):685-93. doi: 10.1016/j.exger.2005.07.007. PMID 16125352
- [Background] Anisimov VN, Egormin PA, Bershtein LM, Zabezhinskii MA, Piskunova TS, Popovich IG, Semenchenko AV. Metformin decelerates aging and development of mammary tumors in HER-2/neu transgenic mice. Bull Exp Biol Med. 2005 Jun;139(6):721-3. doi: 10.1007/s10517-005-0389-9. PMID 16224592
- [Background] Huang X, Wullschleger S, Shpiro N, McGuire VA, Sakamoto K, Woods YL, McBurnie W, Fleming S, Alessi DR. Important role of the LKB1-AMPK pathway in suppressing tumorigenesis in PTEN-deficient mice. Biochem J. 2008 Jun 1;412(2):211-21. doi: 10.1042/BJ20080557. PMID 18387000
- [Background] Nathan DM, Buse JB, Davidson MB, Ferrannini E, Holman RR, Sherwin R, Zinman B; American Diabetes Association; European Association for Study of Diabetes. Medical management of hyperglycemia in type 2 diabetes: a consensus algorithm for the initiation and adjustment of therapy: a consensus statement of the American Diabetes Association and the European Association for the Study of Diabetes. Diabetes Care. 2009 Jan;32(1):193-203. doi: 10.2337/dc08-9025. Epub 2008 Oct 22. PMID 18945920
- [Derived] Kim J, Lim W, Kim EK, Kim MK, Paik NS, Jeong SS, Yoon JH, Park CH, Ahn SH, Kim LS, Han S, Nam SJ, Kang HS, Kim SI, Yoo YB, Jeong J, Kim TH, Kang T, Kim SW, Jung Y, Lee JE, Kim KS, Yu JH, Chae BJ, Jung SY, Kang E, Choi SY, Moon HG, Noh DY, Han W. Phase II randomized trial of neoadjuvant metformin plus letrozole versus placebo plus letrozole for estrogen receptor positive postmenopausal breast cancer (METEOR). BMC Cancer. 2014 Mar 10;14:170. doi: 10.1186/1471-2407-14-170. PMID 24612502